CLINICAL TRIAL: NCT04770493
Title: Proof-of-Concept Clinical Trial of Lamotrigine as a Candidate Pharmacotherapy for Adolescent Alcohol Use Disorder
Brief Title: Enhancing the Effects of Alcohol Treatment With Lamotrigine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004002676; R21AA028394 (NIH)
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol; Teenager; Medication; Clinical Trial
MeSH Terms: conditions — Alcoholism | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lamotrigine (Experimental): Lamotrigine (25 mg/day to 200 mg/day in two divided doses) for 9 weeks
  Interventions: Drug: Lamotrigine
- Placebo (Placebo Comparator): Identical matching placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lamotrigine — Participants will be randomized to lamotrigine (25 mg/day to 200 mg/day in two divided doses) for 9 weeks. A comparator group will receive placebo (sugar pills).
  Other Names: Lamictal
  Arms: Lamotrigine
Drug: Placebo — Matching placebo (sugar pill)
  Arms: Placebo

SUMMARY:
This study will help determine the tolerability and efficacy of the mood-stabilizing anticonvulsant lamotrigine in youth with alcohol use disorder. It will also help establish whether and how lamotrigine improves outcomes related to alcohol use. The results of this proof-of-concept study will inform whether a future larger clinical trial is warranted.

DETAILED DESCRIPTION:
Adolescent alcohol use is a leading public health concern worldwide. Clinical trials have tested a variety of psychosocial interventions with youth that yield only modest short-term benefits. One potential way to improve treatments is to augment psychosocial interventions with pharmacotherapy. The National Institutes of Health has mounted a concerted effort to identify medications that reduce drinking for nearly three decades. Although this effort improved treatment for adults, no medication is indicated for adolescent use and randomized controlled trials with teenagers are almost nonexistent. This gap raises key questions about whether and how medications could benefit youth. Optimizing treatment options for youth requires closing this important gap. Lamotrigine is safe with adolescents and does not adversely interact with alcohol. Lamotrigine targets brain mechanisms implicated in alcohol use disorder, and it has shown to help treat adults with alcohol problems. Yet, despite its widespread use with children and adolescents, no published double-blind, placebo-controlled studies have examined the effects of lamotrigine on drinking-related behavior in youth. The purpose of this study is to determine how well teenagers accept lamotrigine plus alcohol education to reduce adolescent alcohol use. This study will also tell us whether teenagers' alcohol use, craving, and enjoyment of drinking are reduced by lamotrigine.

ELIGIBILITY:
Inclusion Criteria:

* 16 to 24 years old, inclusive
* Self-reports consuming alcohol ≥ 2 days/week on average in the past 90 days of which ≥ 5 days involved ≥ 4 drinks within a 2-hr period (i.e., binge drinking) for boys and ≥ 3 drinks for girls
* Meet the DSM-5 criteria for alcohol use disorder (AUD)
* Be interested in reducing alcohol use
* Be able to read simple English
* Females taking estrogen-containing oral contraceptives have to agree to use secondary methods of birth control, such as condoms because lamotrigine lowers the effectiveness of estrogen-containing oral contraceptives. Sexually active females cannot be in this study if they do not agree to use a barrier method of birth control (condom) every time they engage in sexual intercourse.

Exclusion Criteria:

* Currently receiving formal AUD treatment
* Significant alcohol withdrawal symptoms
* Coexisting moderate or severe substance use disorder other than cannabis and nicotine, as defined by DSM-5 criteria.
* Positive urine toxicology screen any substances other than cannabis (THC)
* Currently taking a pharmacotherapy for AUD, a carbonic anhydrase inhibitor, or a glucuronidation
* Compelled to alcohol treatment by the justice system or has probation or parole requirements that might interfere with study participation
* History of rash that was serious, required hospitalization, or related to lamotrigine
* Have a history of any serious, unstable medical illness including seizures or hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease
* Clinically significant abnormal liver function tests, including elevation of liver enzymes (AST, ALT) 3-fold above the upper limit of normal.
* Abnormal BUN and creatinine for renal impairment
* Renal or hepatic impairment
* Clinically significant abnormalities per physical exam, hematological assessment, bilirubin concentration, or urinalysis
* Pregnant, nursing, or refusing to use a condom, if female.
* Used psychotropic or anticonvulsant medication (prescribed by a health care professional) in the past 30 days (e.g., topiramate)
* Taking medications contraindicated with lamotrigine (e.g., valproate acid [Depakote], carbamazepine, phenytoin, phenobarbital, primidone, and rifampin, protease inhibitors lopinavir/ritonavir and atazanavir/lopinavi
* History of prior treatment with lamotrigine
* Known sensitivity or allergy to lamotrigine
* A previous history of drug reaction with eosinophilia and systemic symptoms (DRESS) or blood dyscrasias
* A history of Steven-Johnson syndrome or any presentation of symptoms suggestive of Steven-Johnson syndrome.
* Current or lifetime history of psychosis or suicidality

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2024-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Miranda, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Per sponsor requirements, all data will be uploaded to the NIAAA Data Repository.
Supporting Information: ICF
Time Frame: One year after the completion of the project.
Access Criteria: As required by the Sponsor, the data from this clinical trial will be uploaded to the National Institute on Alcohol Abuse and Alcoholism (NIAAA) data repository. Like all NIAAA grants, the NIAAA will govern the access criteria.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lamotrigine | Placebo
Started | 23 | 21
Completed | 22 | 19
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lamotrigine | Placebo | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.61 (1.34) | 20.33 (1.43) | 19.95 (1.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 16 | 19 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 12 | 14 | 26
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 44
Drinking Days (%) [Mean (Standard Deviation); unit: Percentage] — Percent of days alcohol was consumed in the past 28 days
  Percentage | 34.32 (11.78) | 37.07 (19.22) | 35.63 (9.98)
Alcohol drinks consumed per drinking day (Mean) [Mean (Standard Deviation); unit: Count of Standard Alcoholic Drinks] — Mean number of standard alcoholic beverages consumed per drinking day in the past 28 days
  Count of Standard Alcoholic Drinks | 4.35 (1.49) | 4.15 (1.55) | 4.25 (1.50)

OUTCOME MEASURES:

1. Primary Outcome: Completion Rates
Description: The number and percentage of youth who complete the active medication phase will determine feasibility.
Time Frame: 9-week active treatment phase
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 23 | 21
Participants | 22 | 19

2. Primary Outcome: Acceptability of the Study Medication
Description: The Client Satisfaction Questionnaire (CSQ-8) ranges from 8 to 32 (higher scores indicate higher satisfaction) and will determine acceptability. Treatment satisfaction will be considered acceptable if the number and percentage of subjects who rate their treatment experience in the "satisfactory" or "highly satisfactory" ranges on the CSQ-8 is equal to or greater than 80%.
Time Frame: 9-week active treatment phase
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 23 | 21
Participants | 20 | 19

3. Secondary Outcome: Alcohol Craving
Description: The primary measure of alcohol craving will be the following single-item: How strong is your craving to drink alcohol? Scores range from 0 (none) to 20 (extremely strong).
Time Frame: 9-week active treatment phase
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 22 | 18
units on a scale | 3.14 (3.41) | 3.81 (4.57)

ADVERSE EVENTS:
Time Frame: 9-week treatment period
Description: Participants are specifically queried each week regarding any adverse events since their last study appointment.
Arm/Group | Lamotrigine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 21/23 | 20/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lamotrigine (N=23) | Placebo (N=21)
Agitation (Psychiatric disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 5 | 1
Loss of Appetite (Metabolism and nutrition disorders) | 3 | 0
Body Aches (General disorders) | 3 | 3
Chills (General disorders) | 2 | 0
Conjunctivitis (Eye disorders) | 1 | 2
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 2 | 5
Fever (General disorders) | 0 | 3
Flu-like symptoms (General disorders) | 5 | 3
Headache (General disorders) | 12 | 5
Sweating (General disorders) | 0 | 2
Hypertension (Cardiac disorders) | 9 | 9
Hypoglycemia (General disorders) | 1 | 4
Impaired Memory (Psychiatric disorders) | 2 | 1
Insomnia (General disorders) | 1 | 1
Irregular Menstruation (Reproductive system and breast disorders) | 1 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Nausea (Gastrointestinal disorders) | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Soar Throat (General disorders) | 5 | 2
Vomiting (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04770493/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/93/NCT04770493/ICF_001.pdf